CLINICAL TRIAL: NCT06848608
Title: Comparison of the Effects of Yoga and Conventional Physiotherapy Programs on Fatigue, Pulmonary Functions and Exercise Capacity in Patients With Sarcoidosis
Brief Title: Comparison of the Effects of Yoga and Conventional Physiotherapy Programs in Sarcoidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Istanbul Saglik Bilimleri University (Other); Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeyda YILDIZ, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYT-2025
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Sarcoidosis; Pulmonary Rehabilitation; Yoga
Keywords: pulmonary rehabilitation; sarcoidosis; yoga
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): The exercises will be taught to the patients one-on-one by the physiotherapist in the hospital. The exercises will be performed 2 days a week for 8 weeks with a group-based, supervised and standardized tele-rehabilitation program and the remaining 3 days of the week with an exercise diary where they will take notes on their continued exercise.
  Program content;
  * Resistance training: Strengthening exercises will be given to the upper and lower extremities
  * Respiratory Training:
  Pursed-lip breathing training Chest breathing exercise Diaphragmatic breathing exercise
  • Thoracic expansion exercises
  In addition, patients in this group will be given free walking 3 days a week in terms of aerobic training.
  Interventions: Procedure: traditional physiotherapy group
- Yoga Group (Active Comparator): The pranayama techniques and asanas in this group will be taught one-on-one by the physiotherapist in the hospital. For 8 weeks, 2 days of the week will be a group-based, supervised and standardized telerehabilitation program, and the remaining 3 days of the week will be followed by an exercise diary in which they will take notes on the continuation of the exercises.
  Content of the program; Pranayamic techniques Asanas
  In addition, patients in this group will be given free walking 3 days a week in terms of aerobic training.
  Interventions: Procedure: yoga program

INTERVENTIONS:
Procedure: traditional physiotherapy group — * Resistance training: It is planned to give strengthening exercises for the upper and lower extremities (quadriceps, hamstrings, gluteus medius, gastrosoleus, deltoids, triceps and biceps brachii) with the resistive exercise band. The fatigue severity perceived by the patients during the exercises is aimed to be 4-6 according to the Modified Borg scale
  * Pursed-lip breathing training (10 repetitions)
  * Chest breathing exercise (10 repetitions)
  * Diaphragmatic breathing exercise (10 repetitions)
  * Thoracic expansion exercises (10 repetitions - apical expansion, unilateral basal expansion, bilateral basal expansion, posterior basal expansion)
  Additionally In terms of aerobic training, free walking will be provided 3 days a week. (Based on distance determined by 6 DYT)
  Arms: Conventional Physiotherapy Group
Procedure: yoga program — Pranayamic techniques:
  Nadi Shodhana: 2 sets of nadi shodhana pranayama consisting of 8 breathing cycles will be applied.
  Ujjai: Two sets of ujjayi technique consisting of 10 breathing cycles with an inhalation:exhalation ratio of 1:2 in each session will be applied with a 1-minute rest period between sets.
  Bhramari: Two sets of bhramari pranayama consisting of 10 breathing cycles will be applied with a low respiratory rate with a 1-minute rest period between sets.
  Sukha Pranayama : It will be applied 5:5 inhalation:exhalation ratio for 5 minutes.
  Kapalabhati: 15 quick breaths in 10 seconds followed by a 20-second break (30 breaths per minute in total) will be practiced for 3 minutes
  Asanas:
  Sukhasana Bharadvajasana Marjaryasana- Bitilasana Bhujaganasana Kapotasana Hasta uttanasana Virabhadrasana I
  In addition, free walking will be given 3 days a week in terms of aerobic training. (Based on distance determined by 6 DYT)
  Arms: Yoga Group

SUMMARY:
Sarcoidosis is a multisystem disease, characterized by the formation of immune granulomas with various clinical symptoms depending on the involved organs, which can involve many organs and systems associated with emotional and physical consequences that affect the quality of life, whose cause is unknown, but usually affects the respiratory system, and occurs mostly in young and middle-aged adults. Lung involvement, seen in 95% of patients, causes limitation of lung capacity and decrease in inspiratory muscle strength, which are important factors that lead to an increase in dyspnea and a decrease in walking distance. In addition to respiratory muscle weakness, skeletal muscle dysfunction is also frequently observed. The most common symptoms in sarcoidosis are dyspnea and fatigue. When the current literature is examined, it can be seen that studies on non-pharmacological treatment methods in Sarcoidosis are quite limited. Although relatively common in Chronic Obstructive Pulmonary Disease (COPD), various studies conducted in patients with Bronchiectasis, Pulmonary Arterial Hypertension and Asthma have shown that yoga results in a decrease in dyspnea and fatigue, and an increase in pulmonary functions and exercise capacity. On the other hand, no study has been found on yogic techniques in Sarcoidosis. Aim of this study is to investigate the effects of yogic techniques and conventional physiotherapy program on pulmonary functions, body oxygen level test (BOLT), exercise capacity (6MWT), anxiety, depression, fatigue, dyspnea perception, sleep quality, and quality of life in sarcoidosis cases at different stages. In these patients known to have multisystem involvement, holistic approaches gain importance due to the nature of the disease.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem disease that can involve many organs and systems, is characterized by the formation of immune granulomas with various clinical symptoms depending on the involved organs, has an unknown cause, but generally affects the respiratory system, and occurs mostly in young and middle-aged adults. Lung involvement, seen in 95% of patients, causes limitation of lung capacity and decrease in inspiratory muscle strength, which are important factors that lead to an increase in dyspnea and a decrease in walking distance. In addition to respiratory muscle weakness, skeletal muscle dysfunction is also frequently observed. The most common symptoms in sarcoidosis are dyspnea and fatigue. Sarcoidosis is a chronic disease associated with emotional and physical consequences that affect quality of life. Psychiatric disorders such as depression and anxiety are more common in patients diagnosed with sarcoidosis than in the general population. Dyspnea, fatigue, respiratory and skeletal muscle weakness observed in patients cause a decrease in quality of life. It is stated that 50% of patients experience sleep disorders and this situation is accompanied by fatigue, anxiety, depression and a decrease in quality of life. The positive effects of exercise training, which is the most important part of multidisciplinary rehabilitation programs in chronic lung diseases, on exercise capacity, dyspnea and fatigue perception, and quality of life in chronic obstructive pulmonary patients have been proven in numerous studies. Respiratory rehabilitation is believed to be an effective treatment method in interstitial lung patients, who often present with restrictive respiratory disorder, due to problems such as increased dyspnea, limitation in exercise capacity, fatigue, anxiety, depression, and low quality of life. This idea is supported by studies showing that pulmonary rehabilitation improves exercise capacity, perception of dyspnea, and quality of life in patients with interstitial lung. Although aerobic and resistance exercise programs are recommended for interstitial lung patients because they increase peripheral muscle strength and tone, the optimal exercise prescription is not yet known. Studies have shown that exercise prescriptions were prepared similarly for COPD patients, and some changes may be required in those with severe disease. Since interstitial lung disease includes many different groups of chronic lung diseases, there is a need for recommendations to consider these different groups in pulmonary rehabilitation practices. Information about the effectiveness of pulmonary rehabilitation programs for sarcoidosis, which is included in the group of interstitial lung diseases, is very limited. According to the guideline published by ERS in 2021, a 6-12 week pulmonary rehabilitation program (at low level of evidence) was recommended for patients with sarcoidosis and fatigue without exercise contraindications to relieve fatigue. It is accepted that the exercise training program applied to sarcoidosis patients provides an increase in exercise capacity and a decrease in fatigue. It has been observed that respiratory exercises applied together with dynamic upper extremity and trunk exercises in young adults provide an improvement in pulmonary functions and it has been stated that these exercises should be added to the treatment program of patients requiring respiratory therapy due to their beneficial effects. Chest wall mobility affects lung functions. Decreased chest wall compliance, especially expansion of the rib cage, leads to atrophy of the diaphragm as well as the intercostal muscles. This can lead to immobility in the thorax, dyspnea and inadequate spontaneous breathing. Thoracic expansion exercises that increase chest wall mobility in individuals with chronic obstructive pulmonary disease have been observed to result in a significant clinical improvement in expired tidal volume, a decrease in dyspnea and an increase in thoracic expansion. Yoga is a combination of asanas, breathing techniques and meditation components and is a suitable approach for cardiopulmonary rehabilitation programs because it regulates autonomic function by increasing vagal nerve activation. Yoga, which increases nitric oxide bioavailability, helps improve endothelial function. Pranayama techniques, which refer to yogic breathing exercises, have been shown to improve pulmonary function in patients with coronary artery disease. Pranayama, which is based on diaphragm techniques, also has positive effects on depression, anxiety, sleep and quality of life. Due to its close connection with the solar plexus, slow and deep breathing activities and asanas performed with diaphragm activation also have beneficial effects in terms of controlling different physical functions and emotional states. Pranayama balances the autonomic nervous system through the tension-related inhibitory stimulations of the nerve endings in the nose and especially the diaphragm. The breathing pattern affects the heart, brain and nervous system and is linked to anxiety. In stressful situations, shorter, more frequent and shallow breathing occurs. The first aim of pranayama is to slow down the respiratory rhythm. Slow and deep breathing reduces stress levels and Partial Arterial Carbon Dioxide Pressure (PaCO2) in the lungs and blood vessels through autonomic reflex stimulation. Parasympathetic nervous system activity is decreased in sarcoidosis patients. During the inspiratory phase of slow pranayamic breathing; "slowly adapting tension receptors" belonging to the lung tissues and sending their signals to dorsal respiratory neurons via the vagal nerve are activated and create inhibitory stimuli in the neural tissue (Hering Breuer reflex). These inhibitory stimuli play an important role in the regulation of airway smooth muscle tone, respiratory pattern, heart rate and systemic vascular resistance. In addition, the tension in the connective tissues around the lungs affects the membrane potential and causes hyperpolarization. Therefore, the inhibitory stimuli and hyperpolarization currents that occur in neural and non-neural tissues as a result of mechanical stretching of the tissues during slow pranayamic breathing exercises lead to modulation of the nervous system and parasympathetic activation. Sarcoidosis patients are generally monitored for a period deemed appropriate by the specialist doctor and do not receive treatment if there is no progression in the disease during this period. Sarcoidosis is mainly treated with cortisone and immunosuppressive drugs that suppress the immune system's response. However, it has been stated that long-term cortisone use can have side effects and can also cause the disease to reoccur. When the current literature is examined, it is seen that studies on non-pharmacological treatment methods in Sarcoidosis are quite limited. Although relatively abundant in COPD, various studies conducted on Bronchiectasis, Pulmonary Arterial Hypertension and Asthma patients have shown that yoga results in a decrease in dyspnea and fatigue, and an increase in pulmonary functions and exercise capacity. On the other hand, no study has been found on yogic techniques in Sarcoidosis. Aim of this study is to investigate the effects of yogic techniques and conventional physiotherapy program on pulmonary functions, body oxygen level test (BOLT), exercise capacity (6MWT), anxiety, depression, fatigue, dyspnea perception, sleep quality and quality of life in sarcoidosis cases at different stages. In addition, holistic approaches gain importance due to the nature of the disease in these patients known to have multisystem involvement, and in this sense, this study is aimed to guide future rehabilitation studies.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Sarcoidosis by a physician (Stage II-III-IV)
* Pulmonary involvement
* Having fatigue symptoms (FAS ≥22 points)
* No immunosuppressive drug use for the last 1 year
* No antidepressant use for the last 6 months

Exclusion Criteria:

* Presence of cognitive impairment that prevents communication
* Anemia
* Uveitis
* Diabetes
* Pregnancy
* Major cardiovascular diseases
* Fractures
* Osteoporosis
* Those who have a neurological or orthopedic disease that will affect the treatment
* Those who are in the exacerbation period of the disease
* Tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Functions | Baseline and week 8
  Spirometric measurement; It will be performed according to ATS/ERS criteria using a spirometer. Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, 25-75% of forced expiratory flow (FEF25-75, forced mid-expiratory flow) and peak expiratory flow (PEF) values can be measured with a spirometer.
Carbon Monoxide Diffusion Capacity of the Lungs (DLCO) | Baseline and week 8
  It measures gas exchange in the lungs. This test evaluates alveolar surface area, membrane integrity and pulmonary capillary blood flow.
Body Oxygen Level Test (BOLT) | Baseline and week 8
  The BOLT result depends on the concentration of carbon dioxide the body can tolerate and the respiratory response to carbon dioxide, and is calculated by breath hold time. It has been stated that BOLT is significantly associated with distance in 6MWT. This provides clinical benefit as it is a cost-free and rapid test as a respiratory function parameter.
Fatigue Assessment | Baseline and week 8
  It is aimed to evaluate fatigue status with the Fatigue Assessment Questionnaire (FAS), which was developed by Michielsen et al. in 2003, is one-dimensional and consists of ten questions and measures physical and psychological fatigue. The total score varies between 10-50. If the FAS score is between 22-34; If you are tired and FAS score is ≥35; is considered overly tired
Exercise Capacity | Baseline and week 8
  A 6-minute walk test is performed for exercise capacity. After resting in a chair for a sufficient period (>30 minutes), patients walk as fast as possible, without running, for 6 minutes on a straight 30-meter corridor. Before and after the test, the patient's fatigue and dyspnea are questioned using the Modified Borg Scale. Oxygen saturation and heart rate are monitored and recorded using a finger pulse oximeter before, during, and after the test.

SECONDARY OUTCOMES:
Respiratory muscle strength measurement | Baseline and week 8
  The patient is seated in a straight-backed chair. After the patient is asked to make a deep exhalation, he is expected to take a deep inspiration for 1-3 seconds. Measurements are repeated 3 times and the highest value is taken.
Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline and week 8
  mMRC is a 0-4 point category scale where patients select the value that best describes their level of dyspnea
Hospital Anxiety and Depression Scale (HADS) | Baseline and week 8
  It includes anxiety and depression subscales. The scale is a self-report scale and consists of a total of 14 items, 7 of which investigate depression and 7 anxiety symptoms. Responses are evaluated in a four-point Likert format and scored between 0-3.
The Pittsburgh Sleep Quality Index | Baseline and week 8
  PSQI consists of 24 questions in total. 19 of these questions are self-evaluation questions. The remaining 5 questions are answered by the individual's roommate or spouse, if any. The first 18 questions answered by the participant are used in calculating the PSQI total score and component scores. The 18 questions answered by the participant provide information on 7 components: sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), use of sleeping pills (component 6), and daytime sleep dysfunction (component 7). Each component is evaluated on a scale of 0-3 points. The sum of these 7 component scores gives the total PSQI score. Total PSQI score varies between 0-21. While the sleep quality of individuals with a total score of 5 or less is considered "good", the sleep quality of individuals with a score above 5 is considered "bad".
Quality of life measured by the St George's Respiratory Questionnaire | Baseline and week 8
  The St George Respiratory Questionnaire (SGRQ) is a standardized questionnaire that measures the effects on general health, quality of daily life and perceived well-being in lung-specific chronic diseases such as chronic obstructive pulmonary disease, asthma, bronchiectasis, kyphoscoliosis, sarcoidosis and cystic fibrosis. It consists of 76 questions in three categories. Its content questions symptoms, activities, and the impact of the disease on daily life. Each section is scored separately between 0-100 points. A score of 0 indicates no impairment in quality of life, while a score of 100 indicates maximum disability and low quality of life. A validity and reliability study of the survey was conducted for the Turkish population.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal D TAKİNACI, PT, Asst Prof, Study Chair — University of Health science
Locations (1):
- Süreyyapaşa Chest Diseases and Chest Surgery Training and Research Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taneja DK. Yoga and health. Indian J Community Med. 2014 Apr;39(2):68-72. doi: 10.4103/0970-0218.132716. PMID 24963220
- [Background] Marcellis RG, Lenssen AF, de Vries J, Drent M. Reduced muscle strength, exercise intolerance and disabling symptoms in sarcoidosis. Curr Opin Pulm Med. 2013 Sep;19(5):524-30. doi: 10.1097/MCP.0b013e328363f563. PMID 23851328
- [Background] Li C, Liu Y, Ji Y, Xie L, Hou Z. Efficacy of yoga training in chronic obstructive pulmonary disease patients: A systematic review and meta-analysis. Complement Ther Clin Pract. 2018 Feb;30:33-37. doi: 10.1016/j.ctcp.2017.11.006. Epub 2017 Nov 11. PMID 29389476
- [Background] Fulambarker A, Farooki B, Kheir F, Copur AS, Srinivasan L, Schultz S. Effect of yoga in chronic obstructive pulmonary disease. Am J Ther. 2012 Mar;19(2):96-100. doi: 10.1097/MJT.0b013e3181f2ab86. PMID 21048431
- [Background] Das RR, Sankar J, Kabra SK. Role of Breathing Exercises in Asthma-Yoga and Pranayama. Indian J Pediatr. 2022 Feb;89(2):174-180. doi: 10.1007/s12098-021-03998-w. Epub 2021 Nov 23. PMID 34812995
- [Background] Baughman RP, Valeyre D, Korsten P, Mathioudakis AG, Wuyts WA, Wells A, Rottoli P, Nunes H, Lower EE, Judson MA, Israel-Biet D, Grutters JC, Drent M, Culver DA, Bonella F, Antoniou K, Martone F, Quadder B, Spitzer G, Nagavci B, Tonia T, Rigau D, Ouellette DR. ERS clinical practice guidelines on treatment of sarcoidosis. Eur Respir J. 2021 Dec 16;58(6):2004079. doi: 10.1183/13993003.04079-2020. Print 2021 Dec. PMID 34140301